CLINICAL TRIAL: NCT07263594
Title: A Phase 1/2, Multicenter, Open-Label, First-in-Human Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Activity of DB-1324 in Participants With Advanced/Metastatic Gastrointestinal Tumors
Brief Title: A Study of DB-1324 in Advanced/Metastatic Gastrointestinal Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: DualityBio Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DB-1324-101
Record Dates: First submitted 2025-11-17; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Gastrointestinal Cancer
Keywords: Gastrointestinal Tumors, DB-1324
MeSH Terms: conditions — Gastrointestinal Neoplasms; Digestive System Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DB-1324 Phase 1 Dose escalation (Experimental): Enrolled Subjects will receive a single-dose of DB-1324 at different Dose Level or different dose regimen
  Interventions: Drug: DB-1324
- DB-1324 Phase 1 Backfill (Experimental): Participants with GI cancers who have received no more than 3 prior lines of systemic therapy may be backfilled at the selected dose regimens to further explore the safety, efficacy, PK, and pharmacodynamics of DB-1324.
  Interventions: Drug: DB-1324
- DB-1324 Phase 1 Dose Expansion (Experimental): Two or more appropriate dose regimens of DB-1324, determined from the emerging dose escalation (and backfill) data, will be explored for preliminary efficacy and safety of DB-1324.
  Interventions: Drug: DB-1324
- DB-1324 Phase 2 (Experimental): Phase 2 will consist of one or more cohorts intended to confirm early signals of efficacy identified in Phase 1.
  Interventions: Drug: DB-1324

INTERVENTIONS:
Drug: DB-1324 — Administered I.V.

SUMMARY:
This study, the first clinical trial, aims to determine the safety, tolerability, pharmacokinetics, pharmacodynamics, maximum tolerated dose, and antitumor activity of DB-1324.

DETAILED DESCRIPTION:
This is a multicenter, open-label, multiple-dose, FIH Phase 1/2 study to explore the safety, tolerability, and efficacy of DB-1324 in participants with malignant GI tumors.

The Phase 1, which includes Dose Escalation, Backfill, and Dose Expansion to identify the MTD and determine the RDEs and RP2D.

Phase 2 will confirm the safety, tolerability, and explore efficacy in selected malignant GI tumors.

For both Phase 1 and Phase 2, participants will receive study treatment until 1) disease progression, 2) loss of clinical benefit in the opinion of the investigator, 3) unacceptable toxicity, 4) withdrawal from study treatment by participant, 5) lost to follow up, or 6) another criterion for discontinuation is met, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically documented advanced/unresectable, or metastatic GI tumor.
2. Have relapsed or progressed on or after standard systemic treatments, or are intolerant to standard treatment, or for which no standard treatment is available.
3. At least one measurable lesion as assessed by the investigator according to response evaluation criteria in RECIST v1.1.
4. Has a life expectancy of ≥ 3 months.
5. Has an ECOG PS of 0-1.
6. Has LVEF ≥ 50% by either ECHO or MUGA within 28 days before enrollment.
7. Has adequate organ functions within 7 days prior to Day 1 of Cycle 1.
8. Has an adequate treatment washout period before Day 1 of Cycle 1.
9. Participants are willing to provide archived tumor tissue or undergo a tumor biopsy for the measurement of CDH17 levels and other biomarkers.
10. Other protocol-defined Inclusion criteria apply.

Exclusion Criteria:

1. Prior treatment with CDH17 targeted therapy.
2. Prior treatment with ADC with topoisomerase I inhibitor.
3. Has chronic enteritis or inflammatory bowel disease. Or has clinically significant bleeding of GI tract or adjacent organs within 1 month prior to the first dose of study treatment. Or has clinically significant obstruction and/or perforation and/or fistulae (including prior GI fistula operation) of GI tract or adjacent tissues within 6 months prior to the first dose of study treatment.
4. Uncontrolled or significant cardiovascular disease.
5. Has a medical history of cerebrovascular accident including transient ischemic attack within 6 months before enrollment.
6. Has a history of (non-infectious) ILD/pneumonitis that required steroids, or has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
7. Have a lung-specific intercurrent clinically significant illness.
8. Has an uncontrolled infection requiring intravenous injection of antibiotics, antivirals, or antifungals.
9. Has clinically active brain metastases.
10. Has unresolved toxicities from previous anticancer therapy.
11. Other protocol-defined Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation and Backfill parts: Percentage of Participants with Dose-Limiting Toxicities (DLTs) as assessed by CTCAE v5.0. | Up to safety follow-up visit, approximately 30 days post-treatment
  Percentage of participants in dose escalation and backfill parts with DLTs
Dose Escalation and Backfill parts: Percentage of Participants with Serious Adverse Events (SAEs) as assessed by CTCAE v5.0. | Up to safety follow-up visit, approximately 30 days post-treatment
  Percentage of participants with SAEs in dose escalation and backfill parts graded according to NCI CTCAE v5.0
Dose Escalation and Backfill parts: Percentage of participants with Treatment Emergent Adverse Events (TEAEs) , Grade ≥ 3 TEAE, TEAE leading to dose reduction/interruption/discontinuation | Up to safety follow-up visit, approximately 30 days post-treatment
  Percentage of participants who experienced any of the above TEAEs in dose escalation and backfill parts graded according to NCI CTCAE v5.0
Dose Escalation and Backfill parts: Maximum Tolerated Dose(MTD) of DB-1324 | Up to safety follow-up visit, approximately 30 days post-treatment
  MTD will be determined by evaluating the incidence of DLTs during the DLT assessment period.

SECONDARY OUTCOMES:
Dose Escalation and Backfill parts: Recommended Dose for Expansions(RDEs) | Up to the completion of Phase 1, assessed up to 12 months
  RDEs will be based on the data collected during dose escalation and backfill parts
Dose Escalation, Backfill and Expansion parts: Recommended Phase 2 Dose(RP2D) | From the beginning of first patient in (FPI) to the end of study, approximately 36 months
  RP2D will be based on the data collected during dose escalation, backfill and expansion parts
Dose Escalation and Backfill parts: Objective Response Rate (ORR) | From the beginning of first patient in (FPI) to the end of study, approximately 36 months
  ORR will be determined by investigator per RECIST v1.1, defined as the percentage of participants who had a best response rating of CR and PR
Dose Escalation and Backfill parts: Duration of Response (DoR) | From the beginning of first patient in (FPI) to the end of study, approximately 36 months
  DoR will be determined by investigator per RECIST v1.1, defined as the time from earliest date of documented CR or PR to the date of documented disease progression or death (by any cause, in the absence of progression)
Dose Escalation and Backfill parts: Disease Control Rate (DCR) | From the beginning of first patient in (FPI) to the end of study, approximately 36 months
  DCR will be determined by investigator per RECIST v1.1, defined as the proportion of participants with best overall response of CR, PR, or SD with confirmation over a period of at least 6 weeks.
Dose Escalation and Backfill parts: Time to Response (TTR) | From the beginning of first patient in (FPI) to the end of study, approximately 36 months
  TTR will be determined by investigator per RECIST v1.1, defined as the time from the first administration to first documented CR or PR.
Dose Escalation and Backfill parts: Progression Free Survival (PFS) | From the beginning of first patient in (FPI) to the end of study, approximately 36 months
  PFS will be determined by investigator per RECIST v1.1, defined as the time from the first administration to documented disease progression or death (by any cause, in the absence of progression), whichever occurs first.
Dose Escalation and Backfill parts: Pharmacokinetic-AUClast | Up to safety follow up visit, approx. 30 days post-treatment
  Area under the concentration-time curve from time 0 to the last of DB-1324, total anti-CDH17 antibody, and unconjugated payload.
Dose Escalation and Backfill parts: Pharmacokinetic-AUC0-τ | Up to safety follow up visit, approx. 30 days post-treatment
  Area under the concentration-time curve from time 0 to time tau of DB-1324, total anti-CDH17 antibody, and unconjugated payload.
Dose Escalation and Backfill parts: Pharmacokinetic-Cmax | Up to safety follow up visit, approx. 30 days post-treatment
  Maximum observed plasma concentration (Cmax) of DB-1324, total anti-CDH17 antibody, and unconjugated payload.
Dose Escalation and Backfill parts: Pharmacokinetic-Tmax | Up to safety follow up visit, approx. 30 days post-treatment
  Time to Cmax of DB-1324, total anti-CDH17 antibody, and unconjugated payload.
Dose Escalation and Backfill parts: Pharmacokinetic-Cthroug | Up to safety follow up visit, approx. 30 days post-treatment
  Trough concentration
Dose Escalation and Backfill parts: Anti-drug antibody (ADA) prevalence | Up to safety follow up visit, approx. 30 days post-treatment
  Percentage of participants who are ADA positive at any point

CONTACTS AND LOCATIONS:
Overall Officials: Lily Hu, Study Director — DualityBio Inc.
Locations (6):
- United States (3):
  - USA02-0, Grand Rapids, Michigan
  - USA01-0, Huntersville, North Carolina
  - USA03-0, Cincinnati, Ohio
- Australia (3):
  - AUS02-0, Randwick, New South Wales
  - AUS03-0, South Brisbane, Queensland
  - AUS01-0, Nedlands, Western Australia